CLINICAL TRIAL: NCT02974582
Title: Understanding How Cigarette Direct Mail Marketing Influence Smoking Behaviors Among High and Low Socioeconomic Status Young Adult Smokers
Brief Title: Understanding How Cigarette Direct Mail Marketing Influences Smoking Behaviors Among High and Low Socioeconomic Status Young Adult Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 170015; 17-MD-0015
Record Dates: First submitted 2016-11-22; First posted 2016-11-28 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-04-17

CONDITIONS: Nicotine Dependence
Keywords: Cigarettes; Behaviors; Attitudes; Beliefs
MeSH Terms: conditions — Tobacco Use Disorder; Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1/Part 1 (Experimental): 60 Participants of high and low SES
  Interventions: Behavioral: Exposure to non health related images
- 2/Part 2 - Discount Coupons (Experimental): Randomized to view direct mail marketing
  Interventions: Behavioral: Exposure to smoking advertising with coupon
- 3/Part 2 - No Discount Coupons (Experimental): Randomized to view direct mail marketing
  Interventions: Behavioral: Exposure to smoking advertising without coupons
- 4/Part 2 - Control (Experimental): Randomized to view direct mail marketing
  Interventions: Behavioral: Exposure to non health related images

INTERVENTIONS:
Behavioral: Exposure to smoking advertising with coupon — Direct mail marketing of smoking advertising with discount coupon
  Arms: 2/Part 2 - Discount Coupons
Behavioral: Exposure to smoking advertising without coupons — Direct mail marketing of smoking advertising without discount coupon
  Arms: 3/Part 2 - No Discount Coupons
Behavioral: Exposure to non health related images — Control group
  Arms: 1/Part 1; 4/Part 2 - Control

SUMMARY:
Background:

Smoking is a major public health problem in the U.S. Almost a half a million Americans die from it in a year. One thing that contributes to why people smoke is the marketing of cigarettes. Cigarette direct mail marketing usually targets young smokers of lower socioeconomic status. Researchers want to find out more about how this kind of marketing influences smoking behavior in young people from different socioeconomic levels.

Objectives:

To study the effects of cigarette direct mail marketing on beliefs, responses, and arousal. To study how these things may differ among young adult smokers of high and low socioeconomic status.

Eligibility:

Volunteer adults ages 18 to 29 who smoke.

Design:

Participants will have 1 visit.

Participants will be asked questions about their health and recent smoking.

A nurse will check their vital signs.

Participants will have a simple eye exam.

They will give blood and urine samples.

Participants will be connected to equipment. This will collect data while they look at pictures.

Then they will have a 10-minute break. A nurse will observe them during the break.

Participants will have their breath analyzed.

Participants will answer questions. The topics will include:

Education

Job

Income

Family history

Tobacco use

Exposure to pro-smoking and anti-smoking messages

History of drug and alcohol use

DETAILED DESCRIPTION:
Smoking remains a public health problem in the US, and cigarette marketing has been concluded as one of the causal factors for the epidemic. Previous studies on cigarette direct mail marketing yielded a limited data on mechanisms influencing smoking behavior. Therefore, there is a need for a study that would provide a stronger evidence on how direct mail marketing influences smoking behavior. The proposed study will consist of two parts where pilot data are to be collected in Part 1, and further data are to be collected in Part 2 conducted as a randomized comparative trial. Up to a total of 530 volunteers ages 18-29 are to be recruited for the study. After meeting the eligibility and enrolling onto the study, participants will have their biospecimens collected followed by an experiment in which they are to be shown images on the computer. Study participants will then take a break and afterwards will provide additional sociodemographic and psychosocial information through an audio computer assisted self-administered interview.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 18 to 29 years, given our focus on young adults.
* Smoking status: Current smokers who report smoking every day and who have smoked at least 100 cigarettes in their lifetime with a breath carbon monoxide level greater than 6ppm per device guidelines
* SES: For the purpose of the study, we will use the empirical groups from our analysis of the Current Population Survey -Tobacco Use Supplement data. Two groups are chosen based on their social determinants and prevalence of smoking.

  1. Low SES: Young adults who do not have a four-year college degree, are not currently enrolled in a four-year college, were born in the US, and have an annual income less than $50,000. This is the group that has been shown to have the highest prevalence of smoking.
  2. High SES: Young adults who are currently enrolled in or graduated from a four year college. This is the group that has been shown to have the lowest prevalence of smoking.
* English proficiency: since study materials are available only in English, only participants who are able to understand English and follow instructions in English are to be enrolled.
* Cognitive ability: Able to understand and willing to sign a written informed consent document.
* General health: Participants need to be generally healthy, as defined as someone with no known significant health problems. Participants can have chronic health conditions if the condition is well managed.

EXCLUSION CRITERIA:

* Inability, in the judgment of the investigator, to understand and follow the requirements of the protocol.
* Currently enrolled in high school.
* Participants with eye conditions that restrict their ability to track an object with their eyes.
* Participants with myopia, hyperopia, and/or astigmatism who cannot pass a simple vision test even with corrective lenses.
* Participants with medical condition(s) that may be triggered by infrared radiation (e.g., epilepsy).
* Self-reported use of alcohol, recreational drugs or prescription medications used for recreational purposes (e.g., amphetamines, cannabis, cocaine, MDMA, ketamines, LSD, opiates and opioids, tranquilizers or opioid analgesics) that may influence their judgement at the time of study in the past 12 hours before the study visit.
* Participants who cannot see an object located between 15 to 27 inches away from them (the required distance between the computer screen and the participants for accurate eye-tracking), even with corrective contact lenses.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 530 (Estimated)
Dates: Start 2026-10-17 (Estimated); Primary Completion 2027-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
To collect pilot data to examine the variability in beliefs, affective responses, and arousal between young adult smokers of high and low socioeconomic status. | 1 Day
  Measure of physiological responses.
To conduct a randomized comparative trial to examine the effect of cigarette direct mail materials on beliefs, affective responses, arousal, and smoking behavior, and their variation by SES among young adult smokers. | 1 Day
  Measure of physiological responses.

SECONDARY OUTCOMES:
To select cigarette direct mail marketing materials that are perceived to be similar in their persuasiveness for Part 2 of the study. | 1 Day
  Measure of physiological responses.

CONTACTS AND LOCATIONS:
Overall Officials: Tsz Chun Choi, Ph.D., Principal Investigator — National Institute on Minority Health and Health Disparities (NIMHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-MD-0015.html